CLINICAL TRIAL: NCT01277913
Title: The Effect of Supplementation With Two Different Doses of Vitamin D (500 IU vs 1000IU)on Bone Mineral Density, Serum 25 Hydroxyvitamin D and Hand Grip Strength in Children With Diabetes Mellitus Type 1 - a Randomized Controlled Trial.
Brief Title: The Effect of Supplementation With Two Different Doses of Vitamin D on Bone Mineral Density, Vitamin D Levels and Hand Grip Strength in Children With Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Dziechciarz, MD, pimiary investigator, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1/2011
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes Mellitus Type 1
Keywords: diabetes; vitamin D; bone density; children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D 1000 IU (Experimental): vitamin D will be given 1000 IU for 12 months
  Interventions: Drug: Vitamin D3
- Vitamin D 500IU (Active Comparator): vitamin D 500 IU will be given for 12 months once daily
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — 1000 IU once daily for 12 months
  Other Names: Vigantoletten 1000
  Arms: Vitamin D 1000 IU
Drug: Vitamin D3 — 500 IU once daily for 12 months
  Other Names: Vigantoletten 500
  Arms: Vitamin D 500IU

SUMMARY:
The aim of the study is to assess the effect of 12 month supplementation with two different doses of vitamin D ( 500 vs 1000) on bone mineral density, serum 25 hydroxyvitamin D levels and hand grip strength in preadolescents with diabetes mellitus type 1.

100 children in the of age 8 -11 with diabetes mellitus type 1 lasting for more than 3 months, without history of diabetic ketoacidosis during previous month, without other chronic disease which may affect calcium-phosphorus metabolism will be randomized in a double blind controlled trial to supplement them with either 500 IU or 1000 IU vitamin D. Every 3 months, in spring summer,autumn and winter serum level of calcium,25-hydroxyvitamin D level and HbA1c will be measured. At the entry and at the end of the study patients will have total body and lumbar spine bone mineral density assessment. Every six months hand grip strength will be measured. Additionally at the beginning and after 12 mo of supplementation and at the beginning serum levels of TNF-alfa, osteoprotegerin and IL-6 will be assessed.

DETAILED DESCRIPTION:
Evidence indicates that majority (75-90%) of children with diabetes have lower serum concentrations of vitamin D, which may negatively impacts bone health and can be associated with reduction of muscular strength. There is still unknown what is the optimal dose of vitamin D in these patients for adequate supply of vitamin D throughout the year to assure optimal peak bone mass and muscle strengthThe aim of the study is to assess the effect of 12 month supplementation with two different doses of vitamin D ( 500 vs 1000) on bone mineral density, serum 25 hydroxyvitamin D levels and hand grip strength in preadolescents with diabetes mellitus type 1.

100 children in the of age 8 -11 with diabetes mellitus type 1 lasting for more than 3 months, without history of diabetic ketoacidosis during previous month, without other chronic disease which may affect calcium-phosphorus metabolism will be randomized in a double blind controlled trial to supplement them with either 500 IU or 1000 IU vitamin D. Every 3 months, in spring summer,autumn and winter serum level of calcium,25-hydroxyvitamin D level and HbA1c will be measured. At the entry and at the end of the study patients will have total body and lumbar spine bone mineral density assessment. Every six months hand grip strength will be measured. Additionally at the beginning and after 12 mo of supplementation and at the beginning serum levels of TNF-alfa, osteoprotegerin and IL-6 will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 8-11 years
* Diabetes type I lasting for more than 3 months
* informed consent given

Exclusion Criteria:

* Adolescence (Tanner stage ≥ 2 for each of the variable)
* Chronic diseases affecting calcium-phosphorus metabolism (hepatic disease, chronic kidney disease, primary phosphate deficiencies, end organ resistance to 1,25OH S genetically)
* Hypervitaminosis D > 200 ng/ml (500 nmol/L)
* Diabetic ketoacidosis during last month

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with normal bone mineral density (z-score>-1)at lumbar spine(L2-L4)and total body after 12mo of supplementation | 12 month
  Bone mineral density will be assessed with DEXA (dual energy X ray absorptiometry)method at the beginning of the study and after 12 month of supplementation with vitamin D
Percentage of patients with adequate 25 hydroxyvitamin level ( >50 ng/ml) | 12 month
  every 3 month in spring summer autumn and winter each patient will have blood testing for the serum level of 25hydroxyvitamin D.
Mean bone mineral density z-score (L2-L4, total body) after 12 mo of supplementation | 12 month
  Bone mineral density will be assessed with DEXA (dual energy X ray absorptiometry)method at the beginning of the study and after 12 month of supplementation with vitamin D
Mean isometric hand grip force | 12 month
  assessed at 6 and 12 mo of supplementation

SECONDARY OUTCOMES:
Mean bone mineral density change after 12 mo of supplementation | 12 mo
Mean serum level of TNF-alfa, osteoprotegerin, IL-6 | 12 mo
Mean HBA1C level | 12 mo
  HBA1c level will be assessed at summer,spring,autumn and winter.
% patients with HbA1C < 7,5 mg% | 12 mo
% patients with vitamin D hypervitaminosis (>200 ng/ml (500 nmol/L) and or hypercalcemia (>2.7 mmol/l) assessed at summer,spring, autumn, and winter | 12 mo
  it will be assessed at summer,spring, autumn, and winter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Warsaw, Poland